CLINICAL TRIAL: NCT01079546
Title: Retrospective Trial to Assess HPV Epidemiology in Squamous Cell Carcinoma of Head and Neck
Brief Title: Human Papillomavirus (HPV) in Squamous Cell Carcinoma of the Head and Neck
Acronym: HPV
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Tel Aviv medical center, Tel Aviv medical center
Other Study IDs: TASMC ZG09 156 CTIL
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-03

CONDITIONS: Epidemiology
Keywords: HPV, Israel, Squamous cell carcinoma of head and neck
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Parafin blocks from squamous cell carcinoma of head and neck
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- Sq.CC of head and neck TASMC
- hadassa Jerusalem
- sheba hospital
- rambam Haifa
- belinson Petah Tikva
- Nazeret
- soroka beer sheva

SUMMARY:
The rationale for this study proposal is derived from previous case series demonstrating that up to 60% of patients with HNSCC, especially in the oropharynx are associated with high risk HPV infection.

In this study, we will characterize the association between HPV infection and HNSCC in Israel and establish a program for its diagnosis and management based on HPV as a biomarker. The rationale for the proposed research is that once it is known which types of HPV are associated with HNSCC, this information can be used to direct diagnosis and screening effort to high risk population. Our approach is based on establishing a multicenter consortium of leading researchers that will establish a joint database of demographic, clinical and biological data from various regions in Israel. For this we have assembled a multidisciplinary research team with the scope and breath (surgical oncology, pathology, virology and molecular biology) needed to complete all phases of the research successfully. The research will be coordinated and performed at the Applied Cancer Research Laboratory, Tel Aviv Sourasky Medical Center. The patients will be recruited from 7 tertiary medical centers in Israel: Ichilov, Bellinson, Hadassa, Rambam, Soroka, Sheba and Nazeret..

DETAILED DESCRIPTION:
To determine the prevalence and classify the high risk human papillomavirus types associated with head and neck cancer in Israel. We will determine the HPV genotype distribution in Israel in order to study the ethnic uniqueness of the region. Many studies have shown HPV 16 to be the most prevalent type in HNSCC (NEJM). In Israeli Jewish women the HPV types 16, 39, 52, and 18 were the most prevalent genotypes found (15). In our aim, we will determine the prevalence of various HPV genotypes in HNSCC specimens.Study population The group will include patients treated with primary surgery or biopsy, with or without adjuvant radiotherapy between 1998 and 2010 for SCC of the oral cavity, oropharynx, hypopharynx, larynx and paranasal sinuses.

The anatomic site and extent of the primary tumor will be documented. The TNM classification of will be based on the staging system revised by the American Joint Committee on Cancer (AJCC). Patients will be recruited from seven national cancer referral hospitals, including Soroka Medical Center in the Negev (Beer Sheva), Sourasky Medical Center (Tel Aviv), Rabin Medical Center (Petach Tikva), Hadassa Medical (Jerusalem), Rambam Medical Center (Haifa), Sheba medical center (Ramat- Gan) and French Hospital Nazareth (Nazareth). These centers cover almost the entire population in Israel, including Israeli Jews, Bedouins, Druze and Israeli Arab population.

Data Entry Data will be entered into a commercially available spreadsheet (Microsoft Excel 2000, Microsoft Corporation, Seattle, WA) and statistical analysis will perform using a computerized software package (SPSS). We have previously used a similar system to report the results of 146 patients with skull base sarcomas in an international multicenter study including 17 cancer centers (17).

Tumor specimens Specimens will be collected retrospectively, and comprise of paraffin sections of primary tumors or biopsies retrived from the pathology department archives at each center. Transportation of paraffin blocks to Tel Aviv for deparaphinization and HPV testing will take place personally by the investigators. Histopathological analysis Primary tumor specimens will be first evaluated by pathologists at each participating cancer. All specimens will be than re-analyzed and evaluated by head and neck pathologist, Dr. Kaplan Ilana. Specimen dissection and tissue sampling of the primary tumor will be in accordance with the current guidelines for the histopathological assessment of head and neck cancer carcinoma.

HPV detection at the laboratory Tissue sections will be subjected to deparaffinization, heatinduced target retrieval, and digestion with proteinase K (Roche Diagnostics, Indianapolis, IN), as described previously (18). DNA is then purified from paraffin by deparaffinization, proteinase K digestion, phenol/chloroform extraction, and ethanol precipitation. We will use the HPV genotyping system using a PCR based HPV GenoArray test kit for genotyping of 37 HPV taypes (Hybribio Limited, Hong Kong). Specimens are placed into PreservCytR LBC medium (ThinPrep liquid Pap vial; Cytyc Corporation). The Amplicor HPV test kit contains a pool of HPV-specific primers designed to amplify HPV DNA from 13 HR genotypes (types 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, and 68). According to the manufacturer's specification, the Amplicor HPV test detects HPV genotypes 31, 52, 58, and 59 at 240 copies/ml and HPV genotypes 16, 18, 33, 35, 39, 45, 51, 56, and 68 at 100 copies/ml with a positivity rate greater than 95%. All genotypes are detected with a 100% positivity rate at 480 copies/ml.

HPV genotyping HPV genotyping is performed by using a commercially available PCR based HPV GenoArray test kit (Hybribio Limited, Hong Kong), which makes use of both DNA amplification and HybriBio's proprietary flowthrough hybridization technique to simultaneously identify 21 HPV genotypes, including 5 low-risk types (types 6, 11, 42, 43, and 44), 14 HR types (types 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68), and 2 intermediate-risk types (types CP8304 and 53).

The test employs a macroarray format with a nylon membrane onto which HPV genotype-specific oligonucleotides probes have been immobilized. In Situ Hybridization system will be performed with Amplicor HPV test (Roche Molecular Systems) for validation of the results. This kit is designed for the detection and discrimination of human papilloma virus (HPV) DNA in paraffinembedded tissue. An HPV16-positive tumor specimen will be used as a positive control.

p16 Immunohistochemistry

The expression status of p16 is strongly correlated with tumor HPV status (19) and therefore we will evaluate the presence of this protein by immunohistochemistry (20). After 5- μ m sections are deparaffinized, antigen retrieval is performed by use of heat-induced epitope retrieval with 10 mM citrate buffer. Immunostaining will be performed with a Ventana automated stainer (Ventana Medical Systems, Tucson, AZ) according to the manufacturer's recommendations. Cervical specimen known to be positive for HPV will be used as positive control and normal tissues as baseline controls. A mouse monoclonal antibody against p16 (MTM Laboratories, Heidelberg, Germany) at 1:500 dilution will be utilized. The p16 antibody is detected using the avidin-biotin-peroxidase technique (Dako LSAB Kit, Dako). On histopathologic review, the pattern of p16 expression is generally dichotomous according to tumor sample, with p16 staining either absent (negative) or present with strong and diffuse nuclear and cytoplasmic staining (positive). Relative protein expression will be estimated using dedicated software (Metamorph, Molecular Devices, Union City, CA), which analyzed the intensity and area of positive staining. Immunohistochemical interpretation will be performed by two investigators blinded to the HPV status and identity of the patient from whom the tumor originated.

Evaluation the association between HPV status and therapeutic response or survival in patients with oropharyngeal/laryngeal SCC Prospective analyses of case series in the United States and Europe have consistently demonstrated that patients with oropharyngeal SCC which are HPV-positive have a better prognosis than patients whose tumors are HPV negative (21,22). We will evaluate the effect of tumor HPV status on treatment response and survival outcomes among patients with oropharyngeal and laryngeal SCC who were treated with primary chemoradiation or radiation therapy (organ preservation regime).

Data Collection Each center will collect data from patients charts. The data will include: age, sex, ethnic group, area of birth and residence, religion, education (ever attendance at school, number of years of school attendance, and age at leaving school), longest occupation, use of tobacco in its different forms, alcohol drinking habits, dietary habits, marital status, sexual history (number of lifetime sexual partners, visits to prostitutes, and frequency of oral sex), histories of various diseases, family history of cancer, and oral cavity health. A "smoker" is defined as an individual who reports having smoked tobacco daily for at least 1 year, and smokers will be asked about duration of smoking and amount and type of tobacco smoked (cigarettes, cigars, pipes or any form of tobacco chewing). A "drinker" is defined as an individual who reports drinking alcoholic beverages at least once a month. Details will be obtained on types of beverages, amounts and duration of habitual drinking. information on tumor-node-metastasis classification and staging will be obtained from the study patients. This classification will be converted into stage according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual. We will evaluate the outcome of each therapy in terms of response (complete response, partial response and progressive disease according to the RECIST classification)

Statistical analysis Five-year overall survival (OS), disease-specific survive al (DSS) and locoregional control rates will be calculated using the Kaplan-Meier method and the difference in survival rate will be assessed by a log rank test (17). OS will be measured from the date of surgery to the date of death or last follow-up. For DSS, the patients who died from causes other than SCC will be censored at the time of death. The variables that will have prognostic potential suggested by univariate analysis will be subjected to multivariate analysis with the Cox proportional hazards regression model. All statistics will be two-sided. A value of P< 0.05 will be considered to indicate statistical significance. Comparison of HPV/p16 classification (three-class model) will be performed by Kruskal-Wallis analysis followed by Wilcoxon rank sum test with Bonferroni corrections. Comparison of protein expression by HPV/p16 classification will be made using one-way analysis of variance (ANOVA) with post hoc comparisons by Dunnett's T3 test. Comparison of HPV - three class model classification status with specific clinical and pathologic variables (sex, TNM stage, T stage, N stage, histologic grade, management, radiotherapy, chemoradiation, alcohol use, tobacco use and clinical response), will be performed by Fisher's exact test. Clinical response will be recorded as complete response versus no response/partial response after completion of treatment. All calculations and analyses will be performed with the Statistical Package for the Social Sciences version 11.5 for Windows (SPSS Inc, Chicago, IL), by a qualified statistician at Tel Aviv Souraky Medical Center (Esther Shabtai PhD).

Sample size and its justification The prevalence of HNSCC in Israel is estimated to be 52 oropharyngeal and 250 laryngeal cancer new cases per year (Middle East cancer consorcium, www.mecc.cancer.gov). The medical centers that will participate in this study cover 80% of the population of the State of Israel. we estimate that the participation rate among case patients will be 89% (range from 76 to 99.0%) (REF JNCI International). Therefore it is estimated a study period of 6 months approximately 100 samples will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* SCC of the oral cavity, oropharynx, hypopharynx, larynx and paranasal sinuses.

Exclusion Criteria:

* pregnancy,
* age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The group will include patients treated with primary surgery or biopsy, with or without adjuvant radiotherapy between 1998 and 2010 for SCC of the oral cavity, oropharynx, hypopharynx, larynx and paranasal sinuses.
  The anatomic site and extent of the primary tumor will be documented. The TNM classification of will be based on the staging system revised by the American Joint Committee on Cancer (AJCC). Patients will be recruited from seven national cancer referral hospitals, including Soroka Medical Center in the Negev (Beer Sheva), Sourasky Medical Center (Tel Aviv), Rabin Medical Center (Petach Tikva), Hadassa Medical (Jerusalem), Rambam Medical Center (Haifa), Sheba medical center (Ramat- Gan) and French Hospital Nazareth (Nazareth). These centers cover almost the entire population in Israel, including Israeli Jews, Bedouins, Druze and Israeli Arab population.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Estimated); Study Completion 2011-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- The Laboratory For Applied Cancer Research, Sourasky Medical Center, Tel Aviv, Israel